CLINICAL TRIAL: NCT06606951
Title: Effect Of Probiotics Supplementation on Outcome Of Malnourished Children Admitted at Assiut University Children's Hospital
Brief Title: Effect Of Probiotics Supplementation on Outcome Of Malnourished Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Gamal Darwish, 71515,Assuit, Assiut University
Other Study IDs: Probiotics Supplementation
Record Dates: First submitted 2024-09-05; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Malnourished Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Outcome Of malnourished children who receive probiotics (Lactobacillus and Bifidobacterium

DETAILED DESCRIPTION:
Acute malnutrition is an imbalance between nutrient requirement and intake, resulting in cumulative deficits of energy, protein, or micronutrients that may negatively affect growth, development, and other relevant outcomes.

Primary acute malnutrition in children is the result of inadequate food supply caused by socioeconomic, and environmental factors, and it is most commonly seen in low- and middle-income countries.

Responsible factors include household food insecurity, poverty, poor nutrition of pregnant women, intrauterine growth restriction, low birth weight, poor breastfeeding and inadequate complementary feeding, frequent infectious illnesses, poor quality of water, hygiene, etc. Therefore, primary acute malnutrition is mostly social rather than biomedical in origin, but it is also multifactorial. The repetitive exposure to pathogens in the environment causes small intestinal bacterial colonization, with accumulation of inflammatory cells in the small intestinal mucosa, damage of intestinal villi, and, consequently, malabsorption of nutrients, which results in malnutrition.

Secondary acute malnutrition is usually due to abnormal nutrient loss, increased energy expenditure, or decreased food intake, frequently in the context of underlying, mostly chronic, diseases like cystic fibrosis, chronic renal failure, chronic liver diseases, childhood malignancies, congenital heart disease, and neuromuscular diseases Acute malnutrition is responsible for almost one third of all deaths in children < 5 years of age and causes intellectual or cognitive impairment among those who survive. he estimated number of underweight children (weight-for-age Z score < -2) globally is 101 million or 16%. In studies using various methods of assessing malnutrition, the prevalence of acute malnutrition among hospitalized children in developed countries ranged from 6 to 51% .

The human gastrointestinal tract harbours microbial populations consisting of 1013-1014 cells . The colonic bacteria are mainly anaerobic and carry out a range of metabolic processes, some of which are considered of benefit to the host. For example, gut microbes ferment indigestible carbohydrates, generating short-chain fatty acids (SCFAs) for the host. These SCFAs have been reported to have several health benefits to the host, including the provision of energy for epithelial cells and lowering the pH of the intestinal lumen, thus restricting growth of some pathogens and providing an anti-inflammatory effect to the host. The gut microbiota has also been observed to play an important role in absorption, storage and expenditure of energy from the diet as well as synthesis of vitamins K and B12 recent studies suggest a link between gut microbiota (GM) and malnutrition with several studies reporting predominance of pathogenic intestinal bacteria in the guts of malnourished children compared to healthy controls. Concordantly, it has been suggested that pathogenic overload leads to persistent enteric inflammation, increased permeability and nutrient malabsorption Such benefits have led to a growing interest in the use of prebiotics, probiotics and other dietary modifications to modulate the gut microbiota to improve nutrition and health Probiotics are defined as "live microorganisms that, when administered in adequate amounts, confer a health benefit on the host For instance, the addition of probiotics to infant formula has been known to confer numerous benefits to the infant, including the improvement of gut health and immunity, countering the growth of harmful bacteria (pathogens) in the gut and enhancing overall host immune and health status

ELIGIBILITY:
Inclusion Criteria:

1- Age group of children from 6 month up to 5 years

Exclusion Criteria:

* age below 6 month and above 5 years

Ages: 5 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The Outcome Of malnourished children who receive probiotics (Lactobacillus and Bifidobacterium)
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Aim of the study | Baseline
  The Outcome Of malnourished children who receive probiotics (Lactobacillus and Bifidobacterium)
perinatal history | Baseline
  1. full term or preterm
  2. type of delivery
  3. NICU admission
Present history | Baseline
  1. disease type
  2. onset
  3. course
  4. duration
  5. stool &urine characters.
Feeding history | Baseline
  1. breast feeding
  2. suckling power
  3. formula feeding
Maternal history | Baseline
  1. The history of pregnancy and delivery
  2. Any maternal complications or illness during the pregnancy
  3. Usage of any drugs
Investigations | Baseline
  1. complete blood count
  2. liver function test
  3. kidney function test
  4. Random blood glucose
Sample size | Baseline
  102 patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sender R, Fuchs S, Milo R. Revised Estimates for the Number of Human and Bacteria Cells in the Body. PLoS Biol. 2016 Aug 19;14(8):e1002533. doi: 10.1371/journal.pbio.1002533. eCollection 2016 Aug. PMID 27541692
- [Result] Bakker GJ, Zhao J, Herrema H, Nieuwdorp M. Gut Microbiota and Energy Expenditure in Health and Obesity. J Clin Gastroenterol. 2015 Nov-Dec;49 Suppl 1:S13-9. doi: 10.1097/MCG.0000000000000363. PMID 26447957
- [Result] van den Elsen LW, Poyntz HC, Weyrich LS, Young W, Forbes-Blom EE. Embracing the gut microbiota: the new frontier for inflammatory and infectious diseases. Clin Transl Immunology. 2017 Jan 20;6(1):e125. doi: 10.1038/cti.2016.91. eCollection 2017 Jan. PMID 28197336